CLINICAL TRIAL: NCT03494699
Title: Effects of App-based Cognitive Training on Cognition in Community Dwelling Elderly Using: A Randomized Controlled Trial
Brief Title: App-based Cognitive Training at Home
Acronym: ACTH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Gangnam Community Health Center (Other); Gangnam-gu Center for Dementia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-02-050
Record Dates: First submitted 2018-02-13; First posted 2018-04-11 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers, Aged

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Multidisciplinary prevention
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Multidisciplinary prevention — group cognitive training (every month) App-based Cognitive Training at Home (using smartphone application) physical activity/body weight/smoking & alcohol cessation monitoring and feedback
  Arms: Intervention group

SUMMARY:
This randomized controlled trial is for investigating the effects of multidisciplinary intervention program on cognition and activity of daily living ability in community dwelling healthy elderly. The intervention consists of cognitive group training every month, daily home cognitive training using cognitive training smartphone application, record of weekly physical activity and body weight and feedback program, and alcohol and smoking cessation monitoring and feedback program. Among these interventions, app-based cognitive training at home is the major intervention in this study. The total duration of intervention is 1 year, and the tablet-based cognitive screening test and the patient-reported questionnaires to evaluate subjective memory decline, quality of life, depression, and activity of daily living are used for outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* literate
* education years >= 6 years
* not demented
* mini-mental status examination >= 24
* android cellular phone users
* no significant decline in activities of daily living (Korea- Instrumental Activities of Daily Living =<5)

Exclusion Criteria:

* Who has a history of major cardiovascular diseases within 3 months of study enrollment (ex. myocardial infarction, stroke)
* Who has current illnesses that could possibly affect cognition or with anticipated life expectancy of less than 2 years (ex. end stage cancer, on chemotherapy)
* Who has a severe hearing difficulty or visual disturbance
* Who has a limitation in communication
* Who was diagnosed with dementia
* Who has a plan for immigration or move in 1.5 years after study enrollment
* Who underwent a cognitive training within 6 months of study enrollment

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-03-22 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Cognition at 6 month | Baseline, 6months
  Table-based cognitive screening test score
Change from Baseline Cognition at 1 year | Baseline, 1year
  Table-based cognitive screening test score

SECONDARY OUTCOMES:
Change in Quality of life measures | Baseline, 6months, 1year
  Quality of life questionnaire
Change in Depression | Baseline, 6months, 1year
  Geriatric depression scale
Change in anxiety | Baseline, 6months, 1year
  Geriatric Anxiety Inventory
Change in Stress | Baseline, 6months, 1year
  Korean version of recognized stress scale
Change in Subjective memory | Baseline, 6months, 1year
  Multifactorial Memory Questionaire
Change in Activities of Daily Living | Baseline, 6months, 1year
  Korean version of Bayer ADL (Bayer Activities of Daily Living)
Change in Dementia Screening Questionnaire score | Baseline, 6months, 1year
  Korean Dementia Screening Questionnaire
Change in Prospective and retrospective memory | Baseline, 6months, 1year
  Prospective and retrospective memory questionnaire
Change in Mastery | Baseline, 6months, 1year
  Mastery questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Dementia Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No